CLINICAL TRIAL: NCT06753201
Title: Prediction of New Regression Equation Using Digital Analysis for Determination of Mesiodistal Width in Permanent Teeth Among a Group of Egyptian Children : a Cross Section Study
Brief Title: Prediction of New Regression Equation Among a Group of Egyptian Children
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Doha Ahmed Ahmed Khalil, dentist, Cairo University
Other Study IDs: mesiodistal dimension of teeth
Record Dates: First submitted 2024-12-22; First posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Regression Equation; Teeth Measurement

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Aim of the study:

Prediction of new regression equation using digital analysis for determination of mesiodistal width of permanent teeth among a group of Egyptian children.

Research question What is the combined mesiodistal dimensions of canines and premolars in a group of 12-15 years old Egyptian children and from it Can the new regression equation predict the size of unerupted canines and premolars?

DETAILED DESCRIPTION:
Tooth size varies significantly between racial groups so mesiodistal dimension in permanent teeth of Egyptian children differ from any international equation, and to the present data, few studies on the mesiodistal dimension of teeth for Egyptian population (Salem et al., 2023).

Tooth size and shape varies from one person to another, from males and females and from one ethnic group to the other depending on genetic factors (Aljuaid et al., 2021).As mandibular incisors are the first teeth to erupt in the permanent teeth and if their dimensions could perhaps be used for predicting the width of unerupted teeth, then it may be advantageous for analysis of mixed dentition at an early age (Moyers, 1976).Environment and genetics both affect tooth size and it's strongly linked to sex and ethnicity. Males' teeth are larger in size than those of the females and Africans have larger teeth than Europeans (Aldeeb, 2021).

Rationale Tooth size differs among and within populations. Tooth size specifically the mesiodistal dimension has an important role in normal occlusion and in arch space analysis as it affects treatment planning and the final results in orthodontic treatment. (Abozeid et al., 2019). Malocclusion is a common esthetic and functional problem in the world. It's a developmental condition caused by alteration in normal development (Ghorbani et al., 2018). The majority of malocclusion, which starts during the mixed dentition period, can be treated and eliminated in its severity if it was managed early (Abozeid et al., 2019).Predicting the size of canines and premolars that have not yet erupted is essential for accurate diagnosis and planning of the optimal course of action throughout the mixed dentition. The exact forecast reveals the difference between the amount of space needed and that which is now available, providing the first component of a successful therapy (Salem et al., 2023)

ELIGIBILITY:
Inclusion Criteria:

- 1. Subjects age between 12-15 years. 2. Positive subjects acceptance for participation in the study. 3. Full set of the permanent dentition from left 1st permanent molar to right 1st permanent molar.

4. Subjects selected with no previous orthodontic treatment to eliminate possibility of any interproximal reduction. 5. Intact marginal ridge

Exclusion Criteria:

- 1. Subjects with history of systemic diseases. 2. Subjects who have any sensitivity or adverse reactions to any of used materials.

3. Subjects with morphologic anomalous.

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study sample will include healthy cooperative children. The children age will range from 12 years to 15 years. They will be selected from the outpatient clinic of Pediatric Dentistry Department of Faculty of Oral and Dental Medicine, Cairo University, according to the following inclusion and exclusion criteria
Sampling Method: Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Measuring mesiodistal width in permanent mandibular anterior teeth, maxillary, mandibular canines and premolars among a group of Egyptian children | baseline
  Measuring mesiodistal width in permanent mandibular anterior teeth, maxillary, mandibular canines and premolars among a group of Egyptian children

SECONDARY OUTCOMES:
New regression equation for determination of mesiodistal width of unerupted canines and premolars. | baseline
  New regression equation for determination of mesiodistal width of unerupted canines and premolars.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Salem, G., Elyazied, M. A., Radwan, E., & Elhiny, O. (2023). New equations for Egyptian children based on Tanaka and Johnston Mixed Dentition Analysis.
- [Background] Abozeid, H., Shiekh, M. E., & AElsayed, M. (2019a). Determination of the Combined Mesiodistal Widths of the Permanent Mandibular Incisors and that of the Maxillary and Mandibular Canines and Premolars in a Group of Egyptian Children in Suez Governorate: A Cross-sectional study.
- [Background] Ling JY, Wong RW. Tanaka-Johnston mixed dentition analysis for southern Chinese in Hong Kong. Angle Orthod. 2006 Jul;76(4):632-6. doi: 10.1043/0003-3219(2006)076[0632:TMDAFS]2.0.CO;2. PMID 16808570